CLINICAL TRIAL: NCT06378190
Title: Multicentre Phase I/IIa Study of Infusion of Autologous Peripheral Blood T Lymphocytes Expanded and Genetically Modified Using Sleeping Beauty Family Transposons to Express a Chimeric Antigenic Receptor With Anti-CD19 Specificity Conjugated to the 4-1BB Co-stimulatory Region and CD3z and huEGFRt Signal Transmission (TranspoCART19) in Patients With Relapsed or Refractory B-cell Lymphoma
Brief Title: Treatment of Relapsed or Refractory B-cell Lymphoma With Chimeric Antigen Receptor (CAR) T-cell Therapy Produced by a New Technology
Acronym: TranspoCART19
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network); Fundación Canaria de Investigación Sanitaria (Other); Fundación para la Investigación Biomédica del Hospital 12 de Octubre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TranspoCART19; 2022-001040-23 (EudraCT Number); 2024-514544-90-00 (EU CTIS Number)
Record Dates: First submitted 2024-02-16; First posted 2024-04-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Refractory B-Cell Lymphoma; B-cell Lymphoma Recurrent
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: Phase I/II, pilot, open, national, prospective, multicentre, non-randomised
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TranspoCART19 cells (Experimental): Adult differentiated, autologous, peripheral blood T lymphocytes, expanded and genetically modified.
  Interventions: Biological: CAR-T cells therapy

INTERVENTIONS:
Biological: CAR-T cells therapy — CAR-T cells therapy

SUMMARY:
The goal of this clinical trial is to to evaluate the safety and efficacy of TranspoCART19 in patients with relapsed/refractory B-lymphoma. The main questions it aims to answer are:

Maximum tolerated dose (MTD) Response rates Participants will be treated with the investigational medicinal product and will be followed for 36 months.

DETAILED DESCRIPTION:
This clinical trial is a Phase I/II, pilot, open-label, national, prospective, multicentre, non-randomised, open-label study to evaluate the safety and efficacy of TranspoCART19 in patients with relapsed/refractory B-lymphoma whose prognosis is less than 2 years.

Phase I: Dose escalation phase with a classic 3+3 design, in which three dose levels of TranspoCART19 will be evaluated: 1 x 106 cells/kg, 3 x106 cells/kg and 5 x 106 cells/kg. The maximum number of patients included in this phase will be 18.

Phase II: an expansion cohort with the maximum tolerated dose (MTD) determined in Phase I.

Patients will be included in the expansion cohort up to a total of 27, including Phase I patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with relapsed or refractory B-cell lymphoma (Diffuse large B-cell lymphoma, Primary diffuse large B-cell lymphoma of the Central Nervous System (CNS), Mantle cell lymphoma, Follicular lymphoma grades 1, 2 or 3a or Marginal lymphoma, including splenic, nodal and MALT).
2. Age over 18 years and under 80 years.
3. Functional status Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1. Patients with ECOG 2 may be included if motivated by haematological disease (Annex 3).
4. Adequate bone marrow haematopoietic reserve.
5. Life expectancy of at least 2 months.
6. Adequate venous access for lymphapheresis. Absence of contraindications for lymphapheresis.
7. Signed informed consent (patient or legal guardian).

Exclusion Criteria:

1. Patients who, in the opinion of a physician, may benefit from other approved potentially curative therapeutic options, including commercial CAR-Ts.
2. Treatment with any experimental or non-commercialised substance in the four weeks prior to recruitment, or who are actively participating in another therapeutic clinical trial.
3. Diagnosis of another neoplasm, past or present. Patients who have been in complete remission for more than 3 years, or with a history of non-melanoma skin cancer or completely resected carcinoma in situ may be included. A current or previous history of clonal T-lymphocytes is also an exclusion criterion.
4. Early relapse after allogeneic haematopoietic stem cell transplantation (less than 3 months for lymphapheresis, less than 6 months for TranspoCART19 infusion) or patients on active immunosuppressive treatment for graft-versus-recipient disease (corticosteroids or other systemic immunosuppressants).
5. Active infection requiring systemic medical treatment.
6. HIV infection.
7. Concurrent and uncontrolled medical illnesses including cardiac, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological or psychiatric illnesses that in the opinion of the investigator pose a risk to the patient.
8. Positive serology for hepatitis B, defined as a positive test for HBsAg. In addition, if the patient is HBsAg negative but has anti-HBcore antibodies, a hepatitis B virus DNA test will be required, and if the result is positive the patient will be excluded.
9. Positive serology for hepatitis C virus (HCV), defined as a positive test for anti-HCV antibodies that is confirmed by Recombinant immunoblot assay (RIBA).
10. Severe organ involvement, defined as cardiac ejection fraction <40%; diffusing capacity of the lungs for carbon monoxide (DLCO) <40%; calculated glomerular filtration rate <30 ml/min; baseline O2 saturation <92%; bilirubin > 2 times upper limit of normal (unless due to Gilbert's syndrome) or transaminases > 2.5 upper limit of normal.
11. Pregnant or lactating women. Women of childbearing age should have a negative pregnancy test at screening.
12. Women of childbearing age, including those whose last menstrual cycle was in the year prior to screening, who are unable or unwilling to use highly effective methods of contraception* from the start of the study until the end of the study.
13. Men who are unable or unwilling to use highly effective methods of contraception* from the start of the study until the end of the study.
14. Need to take glucocorticoids chronically in doses greater than 10 mg/day of prednisone (or equivalent) or other chronic immunosuppressants.
15. Previous anti-CD19 CAR-T therapy. Previous treatment with other anti-CD19 strategies is permitted, provided that CD19 expression has been confirmed in the tumour biopsy.
16. Hypersensitivity to the active substance or to any of the excipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 1 month
  Determine the maximum tolerated dose (MTD) and/or recommended dose of TranspoCART19 cells in patients with relapsed or refractory B-cell lymphoma.
Efficiency | 3 month
  Determine best response rate achieved (overall and complete).

SECONDARY OUTCOMES:
Procedure-related mortality (PRM) | 1 month - 3 month
  Rate of mortality, defined as any death not directly caused by lymphoma.
Toxicity assessment | 1 month - 3 month - 12 month - 36 month
  Number of grade II-IV adverse events using Common Toxicity Criteria (CTC) version 5.0
Response (overall and complete) | 1 month - 3 month - 12 month - 36 month
  Best response rate achieved (overall and complete) following Lugano classification (PET-CT treatment response)
Duration of response | 36 month
  Time (month) in overall response and complete response.
Progression-free survival (PFS) | 12 month - 24 month
  Time (month) between infusion of TranspoCART19 and disease progression or death.
Overall survival (OS) | 12 month - 24 month
  Time (month) between infusion of TranspoCART19 and death of the patient from any cause.
Perceived general well-being | 3 month -6 month -12 month
  Evaluation of quality of life using EuroQol-5 Dimension-5 levels (EQ-5D-5L) questionnaire [score range from 0 (the worst health status for that dimension) to 100 (the best health status)]

OTHER OUTCOMES:
Molecular and cell biology exploratory objectives: Response dynamics | days +28, +100, +180; 9 months - 12 months - 18 months - 24 months - 30 months - 36 month. Biopsy: days 7, 14, 28, 56, 100 and 180 - 6 months - 9 months - 12 months -18 months - 24 months - 36 month.
  Assess disease response dynamics by Positron Emission Tomography (PET)
  - Calculate SUVmax value
Molecular and cell biology exploratory objectives: Response dynamics | days +28, +100, +180; 9 months - 12 months - 18 months - 24 months - 30 months - 36 month. Biopsy: days 7, 14, 28, 56, 100 and 180 - 6 months - 9 months - 12 months -18 months - 24 months - 36 month.
  Assess disease response dynamics by Positron Emission Tomography (PET)
  - Calculate tumour metabolic volume (mL)
Molecular and cell biology exploratory objectives: Response dynamics | days +28, +100, +180; 9 months - 12 months - 18 months - 24 months - 30 months - 36 month. Biopsy: days 7, 14, 28, 56, 100 and 180 - 6 months - 9 months - 12 months -18 months - 24 months - 36 month.
  Assess disease response dynamics by Positron Emission Tomography (PET)
  - Calculate total lesion glycolysis (mL)
Molecular and cell biology exploratory objectives: In vivo survival of TranspoCART19 cells in peripheral blood | 36 month
  Evaluation of time (days) for TranspoCART19 cell survival determined by flow cytometry
Molecular and cell biology exploratory objectives: Analysis of molecular markers which are possibly related to the tumor response to TranspoCART19 cells | Screening and relapse (in case of)
  The tumour biopsy sample obtained prior to infusion of TranspoCART19 cells will be analysed by whole exome study in order to identify possible molecular markers related to the tumor response/resistance to the TranspoCART19 cells.
Molecular and cell biology exploratory objectives: Evaluation of serum biomarkers of toxicity induced by TranspoCART19 cells (cytokine release syndrome and neurotoxicity) | screening, day 0, +1, +7, +14, +21, +28+, 56 and +100.
  Cytokine analyses by ELISA will be performed on the samples collected in order to correlate the obtained data with the development of either cytokine release syndrome or neurotoxicity.
Molecular and cell biology exploratory objectives: Epigenetic studies on mononuclear bone marrow cells. | screening, +28, +100 and relapse (in caso of)
  Epigenomic studies including Conventional and advanced technologies in profiling DNA methylation, histone modifications and ncRNAs.

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital Clínic, Barcelona, Barcelona
  - Institut Català d'Oncologia Hospital, L'Hospitalet de Llobregat, Barcelona
  - Fundación Jiménez Díaz Hospital, Madrid, Madrid
  - Virgen de la Arrixaca University Hospital, El Palmar, Mur
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - University Hospital of Navarra, Pamplona, Navarre
  - Salamanca University Health Care Complex, Salamanca, SALAMANCA
  - Virgen del Rocio Hospital, Seville, Sevilla

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Diez B, Calvino C, Fernandez-Garcia M, Rodriguez-Marquez P, Rodriguez-Diaz S, Martinez-Turillas R, Ceballos C, Illarramendi J, Serrano-Lopez J, Miskey C, Navarro-Bailon A, Lopez-Corral L, Llamas P, Redondo M, Sanchez-Guijo F, Rifon J, Alfonso-Pierola A, Ivics Z, Inoges S, Lopez-Diaz de Cerio A, Yanez R, Bueren JA, Rodriguez-Madoz JR, Prosper F. Generation and GMP scale-up of human CAR-T cells using non-viral Sleeping Beauty transposons for B cell malignances. Mol Ther Methods Clin Dev. 2025 Jan 31;33(1):101425. doi: 10.1016/j.omtm.2025.101425. eCollection 2025 Mar 13. PMID 40034423